CLINICAL TRIAL: NCT05259657
Title: Feasibility, Acceptability, and Preliminary Effects of a Physical Activity Intervention on Psychological Need Satisfaction, Exercise Motivation, Physical Activity Level, and Quality of Life: A Pilot Randomized Controlled Trial Among Young Adult Lymphoma Survivors
Brief Title: Feasibility, Acceptability, and Preliminary Effects of Lymfit
Acronym: Lymfit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Jewish General Hospital (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Christine Maheu, Associate Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MP-05-2021-2560
Record Dates: First submitted 2022-02-08; First posted 2022-02-28 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Cancer Survivors; Lymphoma
Keywords: Cancer survivorship; Quality of Life; Motivation; Physical Activity
MeSH Terms: conditions — Lymphoma; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lymfit intervention (Experimental): Participants randomized to the intervention group will be allocated a pre-registered Inspire II model Fitbit. The kinesiologist will design a personalized exercise prescription for the participant. The kinesiologist will follow up with the participants every 2 weeks for 3 months to discuss their progress and to modify or advance their exercise prescriptions as needed.
  Interventions: Behavioral: Lymfit Intervention
- Wait-list control arm (Other): The control group participants will begin receiving the Lymfit intervention 3 months after they sign the consent form.
  Interventions: Behavioral: Wait-list control

INTERVENTIONS:
Behavioral: Lymfit Intervention — Participants will be allocated a pre-registered Inspire II / Charge IV model Fitbit. The research team will reach out to the participant via videoconferencing and help them to: download the Fitbit smartphone application; log-in using the anonymous study identification information; and pair their Fitbit with their smartphone application.
  A kinesiologist of the study will meet with the participants for a baseline fitness assessment. The kinesiologist will examine the baseline physical activity levels, fitness level and sedentary behaviours of the participants, to design a personalized exercise prescription. Within one week after the baseline fitness assessment, the kinesiologist will contact the participants to discuss the exercise prescription. Every two weeks there-after, the kinesiologist will follow up with the participants via videoconferencing to discuss their progress and to modify or advance their exercise prescriptions as needed, plus an acceptability assessment survey.
  Arms: Lymfit intervention
Behavioral: Wait-list control — Participants will be contacted by the study kinesiologist for a baseline fitness assessment 3 months after they consent, participants will be given a Fitbit, a personalized exercise prescription and receive bi-weekly follow-ups for 12 weeks.
  Arms: Wait-list control arm

SUMMARY:
Background: Lymphoma is one of the most diagnosed cancers in young adults aged 18 to 39. Lymphoma is highly treatable, and the survival rate is often high. Yet, cancer treatments can be toxic, and their side effects can negatively impact the quality of life among cancer survivors. The current research suggests that being active after treatment can improve cancer outcomes. For instance, reducing cancer-related fatigue, anxiety, depression, and improving sleep quality and survival. Physical activities can greatly improve the quality of life after cancer treatment.

Knowledge Gap: Young adults are unique from cancer patients of other age groups. Young adults need stage-of-life-specific, person-centred cancer and survivorship care. Despite knowing that exercise is beneficial in improving cancer outcomes, cancer survivors' engagement and adherence to exercise guidelines remain poor. It is crucial to develop an effective intervention that can motivate lymphoma patients to be active after treatment.

Purposes: Our study team developed a behavioural change intervention named LymFit. The LymFit intervention involves a personalized exercise program, bi-weekly kinesiology follow-ups, and the use of activity trackers. The aim of this study is to test if the design of the intervention is feasible and acceptable. The investigators also aim to test if the intervention is able to promote exercise motivation among young adult lymphoma survivors.

Implications: This 12-week pilot study examines the implementation strategies and clinical relevance of a behavioural change intervention targeting young adult lymphoma survivors. The study results have the potential to map out the optimal design of an effective physical activity intervention in improving cancer outcomes, and optimize post-cancer treatment care coordination among health professionals.

DETAILED DESCRIPTION:
Background: Lymphoma and its subtypes are among the most commonly diagnosed cancers in young adults aged 18 to 39. Most types of lymphoma are often treated with curative therapies. Unfortunately, treatment side effects, and unhealthy or sedentary lifestyles can substantially affect quality of life and long-term cancer prognosis outcomes among young adult cancer survivors.

A growing body of evidence reveals significant associations between physical activity and cancer-related outcomes. Evidence suggests that specific frequency, intensity, timing, and types of physical activity can have positive effects on cancer treatment processes and outcomes. Physical activity is also significantly associated with enhanced health-related quality of life among cancer survivors.

Despite sustained efforts in the development and implementation of exercise interventions geared towards specific cancer populations and age groups, evidence suggests that lymphoma survivors' exercise engagements remain suboptimal. This warrants the development of an intervention that is theoretically guided, and specific to cancer type and age, to enhance physical activity levels sufficient to improve cancer outcomes. Grounded in self-determination theory, the Lymfit intervention (an individualized exercise program with bi-weekly kinesiology assessments and an activity tracker device) supports the psychological need satisfaction of competence, relatedness, and autonomy in engaging physical activities.

Purpose: To evaluate the feasibility, acceptability, and preliminary effects of the Lymfit intervention on participants' motivation to engage in exercise among young adult lymphoma survivors.

Methods: This study is a two-armed feasibility pilot randomized controlled trial. A target sample size of 28 young adult lymphoma survivors (at the end of their treatment up to six months post-treatment) will be randomly allocated to receive either the 12-week Lymfit intervention (intervention group; n=14) or be on a wait-list (control group; n=14). Feasibility will be assessed by examining criteria related to recruitment, randomization, retention, questionnaire completion, and intervention fidelity. Acceptability will be assessed by examining participant satisfaction with the intervention and the perceived suitability of intervention delivery procedures. Preliminary effects will be assessed using self-report questionnaires at baseline and post-intervention with four study outcomes: psychological need satisfaction, exercise motivation, physical activity level, and quality of life.

Implications: This study examines the feasibility and acceptability of the Lymfit intervention. The results of this study are expected to help in mapping out the optimal design of an effective exercise program for improving cancer outcomes and quality of life in young adults with lymphoma. If the Lymfit intervention shows desired effects, it will have to potential to offer nursing professionals an alternative care option to enhance the quality of post-treatment young adults cancer survivorship care.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed lymphoma patients who received an initial diagnosis at the age of 18 to 39
2. Receiving or have received chemotherapy with curative intent within the past six months
3. Own a smartphone that is able to download the Fitbit application
4. Have an internet connection at home that supports participation in coaching sessions via videoconferencing and the ability to complete the study questionnaires online
5. Proficient in either French or English

Exclusion Criteria:

1) Have any contra-indications to moderate to vigorous levels of exercise

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Retention rate from baseline to end of intervention | 3 months
  Measured by calculating the percentage of participants completing the post-intervention survey (retained in the study).
Acceptability of the study procedures assessed using a set of self-report items | 3 months
  10 self-report items examining participant satisfaction with the intervention and perceived suitability of intervention delivery procedures. The items are assessed using a Likert scale ranging from "1. very dissatisfied" to "5. very satisfied".

SECONDARY OUTCOMES:
Change from baseline Psychological Need Satisfaction assessed by The Psychological Need Satisfaction in Exercise (PNSE) scale | 3 months
  The PNSE comprises 18 items and each item is assessed on a six-point Likert scale from false (1) to true (6). There are six items corresponding to each of the three subscales which measure perceived support for competence, autonomy, and relatedness. Subscale scores (ranging from 1 to 6, with higher scores indicating better outcome) are calculated by averaging the scores for the six items that comprise each scale. A mean score of the full scale will also be calculated to represent the overall satisfaction of psychological needs.
Change from baseline Exercise motivation assessed by the Behavioral Regulation in Exercise Questionnaire (BREQ-3) | 3 months
  The multidimensional BREQ-3 instrument comprises 24 items and six subscales each subscale will assess one form of behavioral regulation (i.e., amotivation, external regulation, introjection, identification, integration, and intrinsic regulation). Each question is scored on a five-point Likert scale from not true for me (0) to very true for me (4). The subscales will be weighted to provide an overall estimate of behavioral regulation, the relative autonomy index (RAI), for which higher scores reflect more self-determination.
Change from baseline Exercise level assessed by the Godin-Shephard leisure-time physical activity questionnaire (LTPA-Q) | 3 months
  The LTPA-Q is a 3-item instrument, it asks individuals to recall the number of times in the past seven days they have performed any strenuous, moderate, and mild physical activity of more than 15 minutes in duration.
Change from baseline Quality of life (QoL) assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS-Preference) | 3 months
  The PROMIS-Preference is a 31-item instrument assessing eight domains (29 items) (i.e., anxiety, depression, fatigue, pain interference, physical function, sleep disturbance, ability to participate in social roles and activities, and pain intensity), and Cognitive Function Abilities (2 items). Raw scores generated for each domain are transformed into T scores; higher PROMIS T scores indicate greater endorsement of the construct being assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Publishing study protocol
Supporting Information: Study Protocol
Time Frame: will be submitted to the International Journal of Clinical Trials (IJCT) in March 2022
Access Criteria: Public